CLINICAL TRIAL: NCT07345156
Title: Validation of a Combined Score Combining the Lung Ultrasound Score and Lactate at Discharge for Predicting Early Events After Acute Heart Failure
Brief Title: Congestion and LActate at diScHarge in Acute Heart Failure
Acronym: CLASH-HF
Status: Not yet recruiting | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Other Study IDs: CLASH-HF study
Record Dates: First submitted 2025-12-24; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure Acute; Discharge Follow-up Phone Calls; Mortality Prediction
Keywords: Lung Ultrasound Score; Lactate; Combined score; Acute Heart Failure; Discharge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Integrated LUS-Lactate Risk Group: Patients classified according to a combined assessment of pulmonary congestion measured by lung ultrasound (LUS) and systemic tissue perfusion reflected by blood lactate levels at hospital discharge, aiming to capture both residual congestion and microcirculatory dysfunction and to improve prediction of early adverse outcomes.
  Interventions: Diagnostic Test: Lung Ultrasound Score; Diagnostic Test: Lactate Blood Test

INTERVENTIONS:
Diagnostic Test: Lung Ultrasound Score — A semi-quantitative ultrasound-based measure of pulmonary congestion that estimates interstitial and alveolar edema by counting B-lines across predefined lung zones, providing a simple and reproducible assessment of residual pulmonary congestion in heart failure patients.
Diagnostic Test: Lactate Blood Test — A biochemical marker reflecting the balance between tissue oxygen delivery and consumption, with elevated levels indicating impaired tissue perfusion or increased anaerobic metabolism, and associated with worse outcomes in acute heart failure even in the absence of overt shock.

SUMMARY:
Acute heart failure (AHF) is a leading cause of hospitalization and is associated with high short-term morbidity and mortality, with 20-30% of patients experiencing rehospitalization or death within 30 days. Early adverse events often reflect incomplete recovery, highlighting the need for improved risk stratification after clinical stabilization .Current prognostic approaches mainly focus on hemodynamic congestion. Persistent pulmonary congestion at discharge is a strong predictor of poor outcomes, but these markers primarily assess macrocirculatory abnormalities and do not capture microcirculatory dysfunction, which may persist despite apparent clinical improvement. Lung ultrasound, through the Lung Ultrasound Score (LUS), provides a validated assessment of pulmonary congestion and has demonstrated prognostic value in AHF. However, LUS does not reflect systemic tissue perfusion. In contrast, blood lactate is a robust marker of tissue hypoperfusion, and even mild elevations have been associated with worse outcomes in AHF. A combined score integrating LUS and lactate may therefore better reflect the dual pathophysiology of AHF-persistent congestion and impaired tissue perfusion-and improve prediction of early adverse events.

This protocol aims to validate the prognostic value of this combined score for predicting 30-day rehospitalization or death in patients hospitalized for AHF, with the hypothesis that it outperforms LUS alone.

DETAILED DESCRIPTION:
This is a prospective, multicenter, observational cohort study including adults (≥18 years) hospitalized for acute decompensated heart failure who were deemed clinically stable and scheduled for discharge within 24 hours. Patients with active severe infection or septic shock, significant hypoxemia or respiratory distress requiring advanced oxygen or ventilatory support, advanced liver disease, refusal to participate, or technical inability to perform lung ultrasound were excluded. At discharge, pulmonary congestion was assessed using lung ultrasound with a standardized 8-zone protocol, and venous blood lactate was measured under resting conditions. Demographic data, heart failure phenotype, discharge vital signs, laboratory values, treatments, and hospitalization characteristics were collected. The primary endpoint was a composite of heart failure-related readmission or all-cause mortality within 30 days after discharge. Secondary endpoints included all-cause readmission, emergency department visits at 30 days, and time to first event. Follow-up was conducted at 30 days using a standardized telephone interview and review of medical records, with strict criteria applied for the definition of heart failure readmission.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Hospitalization for acute heart failure/decompensation (clinical diagnosis + imaging/laboratory tests according to local practice).
* Patient deemed ready for discharge (decision made by the team, discharge within 24 hours).

Exclusion Criteria:

* Septic shock/severe active infection at the time of discharge.
* Hypoxemia or respiratory distress requiring high-flow oxygen/ventilation at the scheduled time of discharge.
* Severe cirrhosis/advanced liver failure.
* Refusal to participate.
* Technical impossibility of LUS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Hospitalized for Acute Decompensated Heart Failure:
  Adults admitted due to worsening heart failure symptoms requiring inpatient management, including clinical and/or imaging or laboratory confirmation of decompensation.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Composite of heart failure-related readmission or all-cause mortality | 30 days after hospital discharge
  A combined outcome of heart failure-related rehospitalization or all-cause death within 30 days after hospital discharge, used to assess early adverse events in acute heart failure patients.

SECONDARY OUTCOMES:
Time to first event | At 30 days
  Includes all-cause hospital readmission, emergency department visits within 30 days, and time to the first adverse event, used to evaluate broader short-term outcomes after discharge in acute heart failure patients.

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, Professor, Principal Investigator — LR12SP18 ,University of Monastir
Locations (1):
- Fattouma Bourguiba Hospital of Monastir, Monastir, Monastir Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Núñez J, et al. Lactate and short-term mortality in heart failure. Int J Cardiol. 2019.
- [Background] Rivas-Lasarte M, Alvarez-Garcia J, Fernandez-Martinez J, Maestro A, Lopez-Lopez L, Sole-Gonzalez E, Pirla MJ, Mesado N, Mirabet S, Fluvia P, Brossa V, Sionis A, Roig E, Cinca J. Lung ultrasound-guided treatment in ambulatory patients with heart failure: a randomized controlled clinical trial (LUS-HF study). Eur J Heart Fail. 2019 Dec;21(12):1605-1613. doi: 10.1002/ejhf.1604. Epub 2019 Oct 31. PMID 31667987
- [Background] Gheorghiade M, et al. Congestion in acute heart failure syndromes. Circulation. 2010.
- [Background] Savarese G, Lund LH. Global Public Health Burden of Heart Failure. Card Fail Rev. 2017 Apr;3(1):7-11. doi: 10.15420/cfr.2016:25:2. PMID 28785469
- [Background] Dharmarajan K, Hsieh AF, Lin Z, Bueno H, Ross JS, Horwitz LI, Barreto-Filho JA, Kim N, Bernheim SM, Suter LG, Drye EE, Krumholz HM. Diagnoses and timing of 30-day readmissions after hospitalization for heart failure, acute myocardial infarction, or pneumonia. JAMA. 2013 Jan 23;309(4):355-63. doi: 10.1001/jama.2012.216476. PMID 23340637
- [Background] Gheorghiade M, Vaduganathan M, Fonarow GC, Bonow RO. Rehospitalization for heart failure: problems and perspectives. J Am Coll Cardiol. 2013 Jan 29;61(4):391-403. doi: 10.1016/j.jacc.2012.09.038. Epub 2012 Dec 5. PMID 23219302